CLINICAL TRIAL: NCT01112722
Title: A Multicenter, Randomized, Double Blind, Active Controlled, Parallel Group, Clinical Study, to Evaluate the Safety and Efficacy of Apitox vs Histamine in Subjects With Refractory Osteoarthritis Pain and Inflammation of the Knee
Brief Title: Apitox, Honeybee Toxin for Pain and Inflammation of Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apimeds, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-13
Record Dates: First submitted 2010-04-25; First posted 2010-04-28 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: honeybee toxin; Apitox; pain; inflammation; osteoarthritis; Apitoxin
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Inflammation; Osteoarthritis | interventions — Sodium Chloride; Bee Venoms; Histamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apitox, purified honeybee toxin, injections (Active Comparator): active treatment drug 'Apitox, purified honeybee toxin, lyophilized in saline'
  Interventions: Biological: Apitox, purified honeybee toxin, lyophilized in saline
- histamine injection (Placebo Comparator): the histamine injection produces a similar local effect of pain and erythema as the active drug
  Interventions: Biological: histamine

INTERVENTIONS:
Biological: Apitox, purified honeybee toxin, lyophilized in saline — intradermal injections of 0.1mg apitox in 0.1ml WFI over 12 weeks treatment period, injections twice weekly range from 1 to 20 injections
  Other Names: Apitoxin in Korea
  Arms: Apitox, purified honeybee toxin, injections
Biological: histamine — imitates pain and erythema of honeybee venom
  Arms: histamine injection

SUMMARY:
The study will identify the efficacy of Apitox, purified honeybee toxin, in 330 patients with diagnosed osteoarthritis of the knee. The subjects will be evaluated for relief of pain using Western Ontario and McMaster Osteoarthritis Index (WOMAC) and Physician and Patient Global Assessments and primary efficacy measure of relief of pain and inflammation over a 12 week treatment period after randomization into the trial. Secondary efficacy is improvement of mobility Treatment effect will be compared in a 2-1 Apitox vs active control

DETAILED DESCRIPTION:
feasibility and Site selection has been completed in the US and India

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of one or both knees
* on stable NSAID or none due to intolerance
* women either post menopausal or on stable birth control
* no clinically significant disease or or abnormal laboratory values
* signed informed consent, communicate effectively, understand and comply with all study requirements

Exclusion Criteria:

* serious or unstable medical or psychological condition
* known sensitivity to honeybee venom, histamine or lidocaine
* history of asthma
* any clinically significant ECG abnormalities
* any clinically significant laboratory values OOR
* history of drug or alcohol abuse
* history of joint injury and forms of inflammatory arthritis

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2013-12; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
WOMAC | from 4 wks dose escalation thru 12 weeks treatment dose to 4 wks follow up
  WOMAC

SECONDARY OUTCOMES:
PhGA | from 4 wks global assessment through 12 wks
  physcians global assessment
PGA | from 4 wks throught the 12 wk treatment
  patients global assessmen

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M. H. Kim, M.D., Study Chair — Apimeds, CEO
Locations (14):
- United States (14):
  - Functional Research LLC, Gulf Shores, Alabama
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - SC Clinical Research Inc., Garden Grove, California
  - Axis Clinical Trials, Los Angeles, California
  - Westlake Medical Research, Thousand Oaks, California
  - SC Clinical Research Inc., Upland, California
  - Schrock Orthopedics Research, Fort Lauderdale, Florida
  - AppleMed Research Inc., Miami, Florida
  - Radiant Research Inc., Pinellas Park, Florida
  - Beacon Clinical, Brockton, Massachusetts
  - Radiant Research Inc Columbus, Columbus, Ohio
  - Hillcrest Clinical Research, Olahoma City, Oklahoma
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Tekton Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided